CLINICAL TRIAL: NCT01701141
Title: Depression and Dopamine Transporter Function: A Positron Emission Tomography Study Using C-11 Altropane
Brief Title: Depression and Dopamine Transporter Function Study Using C-11 Altropane
Status: Completed | Type: Observational
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Diego A. Pizzagalli, Associate Professor, Department of Psychiatry, Harvard Medical School, Mclean Hospital
Other Study IDs: 2009-P-001360
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Major Depressive Disorder; Anhedonia
Keywords: Positron Emission Tomography (PET); Magnetic resonance imaging (MRI); reward; stress; learning; Major Depressive Disorder; Anhedonia
MeSH Terms: conditions — Depressive Disorder, Major; Anhedonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Individuals with MDD: Individuals with current MDD as determined by structured clinical interview for DSM-IV (SCID) at time of enrollment.
- Healthy Controls: Individuals with no psychiatric diagnosis as determined by structured clinical interview for DSM-IV (SCID) at time of enrollment

SUMMARY:
Major depressive disorder (MDD) is often characterized by anhedonia and impaired ability to modulate behavior as a function of rewards. However, the neurobiology of anhedonia and reduced reward responsiveness remains largely unknown. Because dopamine (DA) plays a critical role in goal-directed behavior and reinforcement learning, DA dysregulation might play an important role. In fact, several lines of evidence suggest that down-regulation of DA transmission might characterize depression vulnerability and the emergence of depressive symptoms. The current study seeks to elucidate the role of DA dysfunction in MDD. We hypothesize that MDD subjects will show reduced DAT binding potential, reduced reward learning in the probabilistic reward task, and abnormal functional magnetic resonance imaging (fMRI) activation in dorsal and ventral striatal regions during an instrumental learning task.

This study will include three sessions.

The first will take place at Massachusetts General Hospital or at McLean Hospital's Center for Depression, Anxiety and Stress Research. The aims of this session will be to (a) explain the study; (b) collect written informed consent, and (c) assess the subject's eligibility.

Following this, another session (either second or third in order) will take place at the MGH PET Imaging Laboratory. Participants will complete a PET scan and a probabilistic reward task designed to measure reward learning and sensitivity to reward. The radioactive tracer utilized is 11C-altropane.

Another session (either second or third in order) will take place at the McLean Hospital Neuroimaging Center. Participants will complete an instrumental learning task while in the fMRI, followed by a social reinforcement learning task and an implicit learning serial reaction time task upon completion of the scan. In the instrumental learning task, participants have the opportunity to earn money but need to learn, by trial and error, stimulus-outcome associations. The social reinforcement learning task is designed to investigate whether learning deficits in MDD are specific to learning from monetary incentives or whether the learning deficits are more global and are affected when learning from social rewards and punishments. Participants will also complete an implicit learning serial reaction time task, designed to exclude the possibility of global learning deficits in MDD.

ELIGIBILITY:
Criteria for All Subjects

Inclusion Criteria:

1. Written informed consent;
2. Both genders and all ethnic origins, age between 18 and 45;
3. Right-handed (Chapman and Chapman 1987);
4. Absence of any medications for at least 3 weeks;
5. Absence of pregnancy;
6. Absence of current drug use (cocaine, cannabinoids, opiates, amphetamines, benzodiazepines and barbiturates) as assessed by urinary drug test.
7. For women, completion of a negative urine pregnancy test prior to the MRI scan, as well as a negative STAT quantitative serum hCG test immediately prior to radiopharmaceutical exposure;
8. Normal or corrected-to-normal vision and hearing.

Exclusion Criteria

1. Pregnant or currently breast-feeding women or any woman of childbearing potential who is seeking to become pregnant or suspects that she may be pregnant.
2. History or current serious or unstable medical illness, including cancer, cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease;
3. History of seizure disorder;
4. Failure to meet standard PET safety requirements;
5. Failure to meet standard fMRI safety requirements;
6. Students and employees supervised by the Investigators at MGH, McLean Hospital and Harvard University;
7. Absence of fluency in written and spoken English;
8. History of head injury;
9. History or current use of cocaine, stimulants, or other dopaminergic drugs.
10. Diabetes with poor glucose control;
11. History or current diagnosis of dementia, or a score of < 26 on the Mini Mental Status Examination (Folstein, 1975) at the screening visit;
12. Clinical or laboratory evidence of hypothyroidism or currently taking thyroid medication;
13. Currently taking medication that affects blood flow, e.g. certain blood pressure medications
14. Evidence of significant inconsistencies in self-report.

Criteria Specific to MDD subjects

Inclusion Criteria:

1. DSM-IV diagnostic criteria for MDD (diagnosed with the use of the SCID);
2. A baseline HRSD score (Hamilton 1960) greater than or equal to 16 (17-item version);

Exclusion Criteria:

1. Subjects with suicidal ideation where outpatient treatment is determined unsafe by the study clinician. These patients will be immediately referred to appropriate clinical treatment;
2. History or current diagnosis of: learning and developmental disorders (including ADHD and autism spectrum disorders), anorexia nervosa, cognitive disorders, somatoform and factitious disorders, dissociative disorders, personality disorders, organic mental disorders, schizophrenia or other psychotic disorder, bipolar disorder, obsessive compulsive disorder; simple phobia, social anxiety disorder and generalized anxiety disorder are allowed if secondary to MDD.
3. History of substance dependence lifetime or substance abuse within the last 12 months;
4. History of bulimia nervosa or PTSD within the past 2 years;
5. History or current diagnosis of dementia, or a score of < 26 on the Mini Mental Status Examination (Folstein, 1975) at the screening visit;
6. Current use of other psychotropic drugs;
7. Patients with lifetime electroconvulsive therapy (ECT);
8. Presence of any psychotropic medications for at least 2 weeks:

   * 6 months for dopaminergic drugs (including methylphenidate),
   * 6 weeks for fluoxetine,
   * 6 months for neuroleptics,
   * 2 weeks for benzodiazepines,
   * 2 weeks for any other antidepressants.

Criteria Specific to Control subjects

Inclusion Criteria:

1. Absence of medical, neurological, and psychiatric illness (including alcohol and substance abuse), as assessed by subject history and a structured clinical interview (SCID-I/NP);
2. Absence of any medications for at least 3 weeks;

Exclusion Criteria:

1. History or current diagnosis of any of DSM-IV psychiatric illness;
2. First degree relative with mood disorder or psychosis;
3. History or current use of any psychiatric medication.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
11C-Altropane Binding | 1 hour long PET scan during session 2
  11C-altropane binding is recording during the positron emission tomography (PET) scan and is used to measure dopamine transporter levels.
Behavioral Performance in Probabilistic Reward Task | 20 minute task administered during session 2
  The probabilistic reward task is designed to measure sensitivity to reward and reward learning.
Brain Activity during Instrumental Learning Task | 30 minute long fMRI scan during session 3
  Functional magnetic resonance imaging (fMRI) data are acquired while participants perform the instrumental learning task. fMRI data allows us to measure aspects of brain activity.
Behavioral Performance in Instrumental Learning Task | 30 minute task administered during session 3
  The instrumental learning task is designed to measure participant learning from reward and punishment.
Behavioral Performance in the Social Reinforcement Learning Task | 15 minute task administered during session 3
  The social reinforcement learning task is designed to investigate whether learning deficits in MDD are specific to learning from monetary incentives or whether the learning deficits are more global and are affected when learning from social rewards and punishments.

SECONDARY OUTCOMES:
Questionnaire Data | Self-report measures are administered at all 3 sessions which take place within an average of 2-3 weeks
  At all sessions participants will fill out self-report questionnaires regarding aspects of mood and affect, demographics, caffeine and alcohol consumption, etc.
Behavioral Performance in Implicit Learning Serial Reaction Time Task | 5 minute task administered during session 3
  The implicit learning serial reaction time task is designed to exclude the possibility of global learning deficits in major depressive disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Pizzagalli, PhD, Principal Investigator — Mclean Hospital
Locations (2):
- United States (2):
  - McLean Hospital, Belmont, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts